CLINICAL TRIAL: NCT01746732
Title: Effects of Evacetrapib (LY2484595) on the Pharmacokinetics of an Oral Contraceptive in Healthy Female Subjects
Brief Title: A Study of Evacetrapib in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14617; I1V-MC-EIAP (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Moxifloxacin; evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ortho-Cyclen (Experimental): Ortho-Cyclen (35 microgram (mcg) ethinyl estradiol and 250 mcg norgestimate) administered orally, once daily (QD), for 28 days (lead-in period). Then, Ortho-Cyclen orally QD for 28 Days (Days 1 to 28) in one of two treatment periods. Treatment A
  Interventions: Drug: Ortho-Cyclen
- Ortho-Cyclen + Evacetrapib (Experimental): Ortho-Cyclen administered orally, QD, for 28 days (lead-in period). Then, Ortho-Cyclen orally QD for 28 Days (Days 1 to 28) and 130 mg evacetrapib orally, QD, for 21 days (Days 1 to 21) in one of two treatment periods. Treatment B
  Interventions: Drug: Ortho-Cyclen; Drug: Evacetrapib

INTERVENTIONS:
Drug: Ortho-Cyclen — Oral administration
Drug: Evacetrapib — Oral administration
  Other Names: LY2484595
  Arms: Ortho-Cyclen + Evacetrapib

SUMMARY:
The purpose of this study is to evaluate the effects of evacetrapib on oral contraceptives (Ortho-Cyclen®) when given to healthy female participants. The amount of female hormones found in the blood will be measured and compared when taken alone and when taken with evaceptrapib. Each woman will participate in two study periods. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Are pre-menopausal females, and who are healthy as determined by medical history and physical examination
* Have a body mass index of 18 to 30 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Have known allergies to evacetrapib and Ortho-Cyclen (ethinyl estradiol and norgestimate), related compounds or any components of the formulation
* Have a clinically significant abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have taken injectable contraceptives within 12 months prior to the first dose of the lead-in period or topical controlled delivery contraceptives (patch) for 3 months prior to the first dose of the lead-in period
* Use of any tobacco- or nicotine-containing products within 6 months prior to the lead-in phase and during the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ortho-Cyclen: Ortho-Cyclen (OC) of (35 microgram [mcg] ethinyl estradiol and 250 mcg norgestimate) administered orally, once daily (QD) for 28 days (Days 1 to 28)
- Ortho-Cyclen Then Ortho-Cyclen + Evacetrapib; Sequence AB: Treatment A OC administered orally, QD for 28 days (Days 1 to 28)
  Treatment B OC administered orally, QD for 28 days (Days 1 to 28) and 130 milligram (mg) Evacetrapib orally, QD for 21 days (Days 1 to 21)
- Ortho-Cyclen + Evacetrapib Then Ortho-Cyclen; Sequence BA: Treatment B OC administered orally, QD for 28 days (Days 1 to 28) and 130 mg Evacetrapib orally, QD for 21 days (Days 1 to 21)
  Treatment A OC administered orally, QD for 28 days (Days 1 to 28)
Period: Lead-In Period
Arm/Group | Ortho-Cyclen | Ortho-Cyclen Then Ortho-Cyclen + Evacetrapib; Sequence AB | Ortho-Cyclen + Evacetrapib Then Ortho-Cyclen; Sequence BA
Started | 23 | 0 | 0
Participants Received at Least 1 Dose | 22 | 0 | 0
Completed | 22 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Period 1
Arm/Group | Ortho-Cyclen | Ortho-Cyclen Then Ortho-Cyclen + Evacetrapib; Sequence AB | Ortho-Cyclen + Evacetrapib Then Ortho-Cyclen; Sequence BA
Started | 0 | 11 | 11
Completed | 0 | 10 | 11
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Period 2
Arm/Group | Ortho-Cyclen | Ortho-Cyclen Then Ortho-Cyclen + Evacetrapib; Sequence AB | Ortho-Cyclen + Evacetrapib Then Ortho-Cyclen; Sequence BA
Started | 0 | 10 | 11
Completed | 0 | 10 | 7
Not Completed | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Twenty-two subjects received at least one dose of study drug and are included in the summary of subject demographics
Groups:
- Ortho-Cyclen and Ortho-Cyclen + Evacetrapib: Ortho-Cyclen (35 microgram (mcg) ethinyl estradiol and 250 mcg norgestimate) administered orally, QD for 28 days (lead-in period).
  Treatment A Ortho-Cyclen administered orally, QD for 28 Days (Days 1 to 28) Treatment B Ortho-Cyclen orally, QD for 28 Days (Days 1 to 28) and 130 mg evacetrapib orally, QD for 21 days (Days 1 to 21)
Arm/Group | Ortho-Cyclen and Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (6.8)
Sex/Gender, Customized [Number; unit: Participants]
  Females | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 11
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Ethinyl Estradiol
Time Frame: Day 21: Predose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16 and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/ml)
Groups:
- Ortho-Cyclen: Ortho-Cyclen (35 microgram (mcg) ethinyl estradiol and 250 mcg norgestimate) administered orally, once daily (QD), for 28 days (lead-in period). Then, Ortho-Cyclen orally QD for 28 Days (Days 1 to 28) in one of two treatment periods.
  Ortho-Cyclen: Oral administration
- Ortho-Cyclen + Evacetrapib: Ortho-Cyclen administered orally, once daily (QD) for 28 days (Days 1 to 28) and 130 mg Evacetrapib orally, once daily (QD) for 21 days (Days 1 to 21)
Arm/Group | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 16 | 17
picogram per milliliter (pg/ml) | 71.7 (35) | 70.6 (37)

2. Primary Outcome: PK: Area Under the Concentration Curve Over a 24 Hour Dosing Interval (AUCτ) of Ethinyl Estradiol
Time Frame: Day 21: Predose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16 and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram x hour per ml (pg*hour/ml)
Groups:
- Ortho-Cyclen + Evacetrapib: Ortho-Cyclen administered orally, QD, for 28 days (lead-in period). Then, Ortho-Cyclen orally QD for 28 Days (Days 1 to 28) and 130 mg evacetrapib orally, QD, for 21 days (Days 1 to 21) in one of two treatment periods.
  Ortho-Cyclen: Oral administration Evacetrapib: Oral administration
Arm/Group | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 16 | 17
picogram x hour per ml (pg*hour/ml) | 907 (31) | 840 (28)

3. Primary Outcome: PK: Minimum Observed Drug Concentration (Cmin) of Ethinyl Estradiol
Time Frame: Day 21: Predose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16 and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Arm/Group | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 16 | 17
pg/ml | 15.9 (65) | 13.2 (66)

4. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Ethinyl Estradiol
Time Frame: Day 21: Predose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16 and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hour
Arm/Group | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 16 | 17
hour | 3.00 [0.50 to 12.00] | 4.00 [1.02 to 5.00]

5. Primary Outcome: PK: Maximum Concentration (Cmax) of Norelgestromin
Time Frame: Day 21: Predose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16 and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Arm/Group | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 16 | 17
pg/ml | 1410 (21) | 1830 (17)

6. Primary Outcome: PK: Area Under the Concentration Curve Over a 24 Hour Dosing Interval (AUCτ) of Norelgestromin
Time Frame: Day 21: Predose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16 and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hour/ml
Arm/Group | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 16 | 17
pg*hour/ml | 16200 (21) | 18100 (22)

7. Primary Outcome: PK: Minimum Observed Drug Concentration (Cmin) of Norelgestromin
Time Frame: Day 21: Predose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16 and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Arm/Group | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 16 | 17
pg/ml | 397 (35) | 422 (34)

8. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Norelgestromin
Time Frame: Day 21: Predose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16 and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hour
Arm/Group | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Number analyzed (Participants) | 16 | 17
hour | 3.53 [2.00 to 12.00] | 4.00 [1.02 to 5.00]

ADVERSE EVENTS:
Groups:
- Ortho-Cyclen (Lead-in Phase): Ortho-Cyclen oral doses of (35 mcg ethinyl estradiol and 250 mcg norgestimate) once daily for 28 days (Days 1 to 28)
- Ortho-Cyclen: Ortho-Cyclen (35 microgram (mcg) ethinyl estradiol and 250 mcg norgestimate) administered orally, once daily for 28 days (lead-in period). Then, Ortho-Cyclen orally for 28 Days (Days 1 to 28) in one of two treatment periods.
  Ortho-Cyclen: Oral administration
- Ortho-Cyclen + Evacetrapib: Ortho-Cyclen administered orally for 28 days (lead-in period). Then, Ortho-Cyclen orally for 28 Days (Days 1 to 28) and 130 mg evacetrapib orally for 21 days (Days 1 to 21) in one of two treatment periods.
  Ortho-Cyclen: Oral administration
  Evacetrapib: Oral administration
Arm/Group | Ortho-Cyclen (Lead-in Phase) | Ortho-Cyclen | Ortho-Cyclen + Evacetrapib
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/17 | 0/21
Other Adverse Events (participants affected / at risk) | 9/22 | 5/17 | 5/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ortho-Cyclen (Lead-in Phase) (N=22) | Ortho-Cyclen (N=17) | Ortho-Cyclen + Evacetrapib (N=21)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 1 (1) | 5 (5)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days